CLINICAL TRIAL: NCT03142763
Title: Assessment of TMAO Formation With Egg Intake Versus Choline Supplement in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Maria Luz Fernandez, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H16-194
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Eggs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg intake (Experimental): Consumption of 3 eggs per day for breakfast, 4 weeks
  Interventions: Other: Eggs
- Choline Supplement intake (Experimental): Consumption of choline supplement, 1 1/2 tablet (395mg choline), with breakfast for 4 weeks
  Interventions: Dietary Supplement: Choline Supplement

INTERVENTIONS:
Other: Eggs — Consumption of 3 eggs per day for breakfast, 4 weeks
  Arms: Egg intake
Dietary Supplement: Choline Supplement — Consumption of choline supplement, 1 1/2 tablet (395mg choline), with breakfast for 4 weeks
  Arms: Choline Supplement intake

SUMMARY:
The objective of this study is to determine the effects of consuming either 3 eggs per day as compared to a daily choline supplement (choline bitartrate, 397.5 mg choline/day) on plasma concentrations of High Density Lipoprotein-cholesterol (HDL-C), trimethylamine N-oxide (TMAO), and other biomarkers of cardiovascular disease risk in young, healthy individuals. The goal is to determine if choline given as phosphatidylcholine (eggs) will lead to a different TMAO response when compared to choline in free supplemental form.

DETAILED DESCRIPTION:
Epidemiological data in short term studies, suggests that egg intake does not increase risk for cardiovascular disease (CVD). In fact, eggs are a great source of phospholipids (phosphatidylcholine) where choline has many metabolic roles, specially in lipid metabolism and cell membrane structure. Choline is present in the diet as free choline, which is absorbed in the small intestines, or choline esters, which is absorbed intact primarily through the lymphatic system. In addition, recent evidence suggests that the choline found in eggs may be metabolized by intestinal microbes into trimethylamine N-oxide (TMAO), a compound that may increase the risk for CVD. However, it is not known to what extent egg intake may contribute to plasma TMAO concentrations.

Therefore, the objective of this study is to determine the impacts of daily intake of 3 eggs versus a choline supplement on plasma TMAO as well as other biomarkers for CVD risk, with the goal of determining if the same amount of choline given as phosphatidylcholine from eggs will increase plasma choline levels without a concomitant increase in plasma TMAO, such that CVD risk is not negatively impacted.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (18-30 years), BMI 18.5 - 29.9 kg/m2, proficient in English, and willing to consume 3 eggs per day or 397.5 mg of choline supplement (1½ tablets/day) for 4 weeks each.

Exclusion Criteria:

* Self-reported diabetes mellitus, cardiovascular disease, history of stroke, renal problems, liver disease, cancer, or a diagnosed eating disorder
* Taking any glucose-lowering prescriptions or supplements, triglyceride-lowering medications, bile acid sequestrants, or high dose chromium or cinnamon supplements
* Taken antibiotics in the previous 1 months, or if they are vegetarian or vegan
* BMI ≤ 18.4 or ≥ 30 kg/m2, or extreme clinical values, such as plasma triglycerides > 500 mg/dL, plasma glucose > 126 mg/dL, plasma cholesterol > 240 mg/dL, plasma creatinine ≤ 0.5 or ≥ 0.9 mg/dL for females and ≤ 0.7 or ≥ 1.2 mg/dL for males, or blood pressure > 140/90 mm Hg (average of 3 readings)
* Allergic to eggs or any component of the choline supplement

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Eggs of Egg Consumption on Plasma Biochemical Parameters | 1 year
  Using plasma form each participant, an automated spectrophotometer is able to analyze at once plasma lipids [total colesterol, triglycerides, HDL (mg/dL)], glucose (mg/dL), CRP (mg/dL, and liver enzymes [alanine aminotransferase and aspartate aminotransferase (U/L)].

SECONDARY OUTCOMES:
Effects of Intervention on Gene Expression using RT-PCR | 1 year
  PBMC will be isolated from whole blood. RNA will be isolated from these cells, and then cDNA will be synthesized using a specific kit. Finally a RT-PCR will be used to analyze the expression of genes, such as: GAPDH, HMG-CoA reductase, LDL-r, CD36, SRA, FMO3, SRB1, PPAR-gama. All results will be presented based on house keeping gene GAPDH.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luz Fernandez, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No